CLINICAL TRIAL: NCT06805487
Title: A Phase 1 Evaluation of the Protective Efficacy of a Single Dose of the Live Attenuated Tetravalent Dengue Vaccine TV003 or Previous Zika Infection Against Infection With ZIKV-SJRP Challenge Compared to DENV and ZIKV-naïve Historical Controls Against Infection With ZIKV-SJRP Challenge
Brief Title: Evaluation of the Protective Efficacy of TV003 or Previous Zika Infection Against Infection With ZIKV-SJRP Challenge Compared to DENV and ZIKV-naïve Controls Against Infection With ZIKV-SJRP Challenge
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: Johns Hopkins Bloomberg School of Public Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: CIR 369
Record Dates: First submitted 2025-01-28; First posted 2025-02-03 (Actual); Last update posted 2025-02-03 (Actual); Status verified 2025-01

CONDITIONS: Zika Virus
MeSH Terms: conditions — Zika Virus Infection | interventions — Plasmalyte A

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Arm 1: DENV/ZIKV naive subjects receiving TV003 (Experimental): Twelve volunteers will receive TV003 followed by challenge with ZIKV on Day 180 (6 months post-vaccination).
  Interventions: Biological: TetraVax-DV-TV003 (TV003); Biological: Challenge virus ZIKV-SJRP/2016-184
- Infectivity Controls: DENV/ZIKV naive subjects receiving PlasmaLyte (Placebo Comparator): Four volunteers will receive PlasmaLyte as control followed by challenge with ZIKV at least 28 days after vaccination.
  Interventions: Biological: Plasmalyte; Biological: Challenge virus ZIKV-SJRP/2016-184
- Arm 2: Subjects with previous ZIKV infection (Experimental): Previous ZIKV-infected volunteers will be challenged with ZIKV on Arm 2 Day 0.
  Interventions: Biological: Challenge virus ZIKV-SJRP/2016-184

INTERVENTIONS:
Biological: TetraVax-DV-TV003 (TV003) — 0.5 ml of TV003 delivered via subcutaneous injection. TV003 contains 10^3.3 plaque forming units (PFU)/mL of rDEN1Δ30, 10^3.3 PFU/mL of rDEN2/4Δ30(ME), 10^3.3 PFU/mL of rDEN3Δ30/31- 7164 and 10^3.3 PFU/mL of rDEN4Δ30
  Arms: Arm 1: DENV/ZIKV naive subjects receiving TV003
Biological: Plasmalyte — 0.5 mL of PlasmaLyte delivered via subcutaneous injection
  Arms: Infectivity Controls: DENV/ZIKV naive subjects receiving PlasmaLyte
Biological: Challenge virus ZIKV-SJRP/2016-184 — 0.5 ml of ZIKV-SJRP/2016-184 delivered via subcutaneous injection. ZIKV-SJRP/2016-184 contains a dose of 10^2 plaque-forming units (PFU).

SUMMARY:
Zika virus (ZIKV) is an illness people can get from mosquitoes. The infection is generally mild with symptoms that include a fever, rash, red eyes, and joint pain, though most of those infected have no symptoms. Preventing ZIKV is important because if a pregnant person is infected with ZIKV, it can cause birth defects in their unborn child.

The goals of this study are to find out if people who have already been infected with one type of ZIKV can get infected with ZIKV a second time, and to test the ability of the TV003 dengue vaccine to prevent people from getting infected with the ZIKV-SJRP challenge virus.

DETAILED DESCRIPTION:
This study is an open label with 2 study arms. Arm 1 will evaluate the protective efficacy of TV003 against ZIKV challenge. Arm 1 will include infectivity controls who will receive PlasmaLyte (the TV003 diluent) and the treatment assignment will be blinded to reduce bias in the assessment of adverse events. The PlasmaLyte recipients will serve as infectivity controls to ensure the potency of the ZIKV challenge. The treatment assignment of the infectivity controls may be unblinded as early as 28 days after receipt of TV003/PlasmaLyte if they are needed for ZIKV-challenge of volunteers in Arm 2 and may be challenged earlier than the TV003 cohort. Arm 2 will evaluate the protective efficacy of previous ZIKV infection against subsequent ZIKV challenge. Both arms will be compared to historical controls who previously received ZIKV infection. Infectivity controls will not be included in the efficacy analysis.

This study will include 16 flavivirus-naïve subjects for Arm 1. Twelve subjects will receive the live attenuated dengue vaccine candidate TV003 at Study Day 0 and 4 subjects will receive PlasmaLyte at Study Day 0. These subjects will be randomized in blocks of 4 (3 TV003:1 PlasmaLyte). At Study Day 180, Arm 1 subjects will receive the controlled human infection strain of ZIKV SJRP/2016-184 as a challenge virus. These subjects will include those volunteers who received TV003 and at least 1 of the infectivity controls who received PlasmaLyte. Subjects in Arm 1 will be followed for approximately 52 weeks (approximately 360 days) from the time of vaccination.

Ten subjects who had a ZIKV infection, either from a previous ZIKV controlled human infection study where they had received either ZIKV SJRP/2016-184 or ZIKV Nicaragua/2016 or were excluded during screening for previous studies as having ZIKV infection, will be enrolled as a group in Arm 2. Subjects enrolled in Arm 2 will be challenged with the ZIKV SJRP/2016-184 challenge virus separately from TV003 recipients. At least 1 of the PlasmaLyte recipients enrolled in Arm 1 on Day 0 will be included in this group to receive ZIKV SJRP/2016-184 as an infectivity control. Arm 2 subjects will be followed after ZIKV challenge for approximately 26 weeks (approximately 180 days). Subjects will be screened for eligibility up to 60 days prior to vaccination on Study Day 0.

ELIGIBILITY:
Inclusion Criteria:

* Adults between 18 and 40 years of age, inclusive.
* Good general health as determined by physical examination, laboratory screening, and review of medical history.
* Available for the duration of the study, approximately 52 weeks.
* Willingness to participate in the study as evidenced by signing the informed consent document.
* Must be able to complete the informed consent process and comprehension assessment independently and without assistance.
* Subjects assigned male at birth: Willingness to use barrier contraception during cervico-vaginal, anal, and oral intercourse from Study Day 0 through 90 days post ZIKV challenge (in accordance with CDC guidance).
* Subjects assigned female at birth: Willingness to use barrier contraception during cervico-vaginal, anal, and oral intercourse from Study Day 0 through 56 days post ZIKV challenge (in accordance with CDC guidance).
* Subjects of childbearing potential must be willing to use effective contraception through 56 days post-ZIKV challenge, in accordance with CDC guidance. Reliable methods of contraception include hormonal birth control* (implantable, hormonal patch, hormonal vaginal ring, oral contraception, Depo-Provera injection, etc.), surgical sterilization (hysterectomy, tubal ligation, or tubal coil at least 3 months prior to inoculation with TV003/PlasmaLyte and/or ZIKV challenge), and intrauterine device. All subjects assigned female at birth will be considered having child-bearing potential except for those with post-menopausal status documented as at least 1 year since last menstrual period, those assigned female at birth who have sex with partners assigned female at birth (exclusively) and have no intention of conceiving a child during the study, and for the vaccination phase of the study only, participants who practice abstinence (≥ 6 months with no sexual contact). Subjects who are not considered to be of childbearing potential will not be required to use contraception other than barrier contraception for the purpose of reducing potential transmission.

  * Volunteers on hormonal birth control must not be on medications or other agents that decrease the effectiveness of hormonal birth control.

Inclusion Criteria for Challenge with ZIKV SJRP/2016-184:

* Currently enrolled in the study.
* Good general health as determined by physical examination and review of medical history.
* Available for the duration of the study, which is approximately 26 weeks after challenge.
* If the challenge portion of the study is expected to begin from March 16-October 30, subject is willing to reside in the inpatient unit for 6 days (or longer for safety if necessary) following receipt of ZIKV.
* Willingness to participate in the study as evidenced by signing the informed consent document.
* Female assigned at birth only: Female assigned at birth subjects of childbearing potential should be willing to use highly effective contraception for the duration of the trial. Reliable methods of contraception include hormonal birth control, surgical sterilization, and intrauterine device. All female assigned at birth subjects will be considered as having childbearing potential in this phase of the study, except for those who have had a hysterectomy, tubal ligation, or tubal coil (at least 3 months prior to vaccination), or who are considered to be post-menopausal, as documented by at least 1 year since last menstrual period.

Additional Inclusion Criteria for Arm 2 Subjects with a Previous History of ZIKV Infection Only:

-History or serologic evidence of previous ZIKV or identified as an infectivity control.

Exclusion Criteria:

* Currently pregnant, as determined by positive beta-human choriogonadotropin (b-hCG) test, breast-feeding, planning to become pregnant during the 12-month duration of the study or planning to donate eggs through 56 days post ZIKV challenge. A careful detailed reproductive and contraception use history will be obtained and the subject will be excluded if the history or clinical record raises concerns related to pregnancy prevention.
* Evidence of clinically significant neurologic, cardiac, pulmonary, hepatic, rheumatologic, autoimmune, or renal disease by history, physical examination, and/or laboratory studies.
* Behavioral, cognitive, or psychiatric disease that in the opinion of the investigator affects the ability of the subject to understand and cooperate with the requirements of the study protocol.
* Evidence of recent opiate use based on urine toxicology screen.
* Screening laboratory values of Grade 1 or above for absolute neutrophil count (ANC), ALT, and serum creatinine, as defined in this protocol.
* Any other condition that in the opinion of the investigator would jeopardize the safety or rights of a subject participating in the trial or would render the subject unable to comply with the protocol.
* Any significant alcohol or drug abuse in the past 12 months which has caused medical, occupational, or family problems, as indicated by subject history.
* History of a severe allergic reaction or anaphylaxis.
* Severe asthma (emergency room visit or hospitalization within the last 6 months).
* HIV infection, by screening and confirmatory assays.
* Hepatitis C virus (HCV) infection, by screening and confirmatory assays.
* Hepatitis B virus (HBV) infection, by Hepatitis B surface antigen (HBsAg) screening.
* History of Guillain-Barré syndrome (GBS).
* History of seizure disease or peripheral neuropathy.
* History of any neuroinflammatory disorder, i.e., Bell's Palsy, transverse myelitis.
* Any known immunodeficiency syndrome, including that caused by malignancy.
* Use of anticoagulant medications, (use of antiplatelet medication such as aspirin or non-steroidal anti-inflammatory medication is permitted and will not exclude a subject from enrollment).
* Use of corticosteroids (excluding topical, inhaled, or nasal) or immunosuppressive drugs within 28 days prior to or following vaccination. Immunosuppressive dose of corticosteroids is defined as ≥10 mg prednisone equivalent per day for ≥14 days.
* Receipt of a live vaccine within 28 days or an inactivated or subprotein vaccine within the 14 days prior to vaccination or anticipated receipt of any vaccine during the 28 days following vaccination with the exception of the inactivated influenza vaccine and COVID 19 vaccines either licensed or under EUA which can be given at any time, however all effort will be made to avoid giving influenza and COVID-19 vaccines within the above windows.
* Asplenia.
* Receipt of blood products within the past 6 months, including transfusions or immunoglobulin or anticipated receipt of any blood products or immunoglobulin during the 28 days following vaccination.
* Anticipated receipt of any investigational agent in the 28 days before or after vaccination.
* Subject has definite plans to travel to a ZIKV endemic or dengue endemic area during the study.
* Previous hypersensitivity to any study product component.
* Refusal to allow storage of specimens for future research.
* Subject is a JHU student currently enrolled in a coursework, an internship, or clinical hours where the supervisor or instructor of record is employed by the Center.
* Subject is faculty or staff currently employed by the Center.

Additional Exclusion Criteria for TV003/PlasmaLyte Group Only:

* History or serologic evidence of previous ZIKV, dengue virus infection, yellow fever virus, St. Louis encephalitis virus, or West Nile virus.
* Previous receipt of a flavivirus vaccine (licensed or experimental).

Exclusion Criteria for ZIKV SJRP/2016-184:

* Female assigned at birth only: Currently pregnant, as determined by positive B- HCG test, or breast-feeding.
* Evidence of clinically significant neurologic, cardiac, pulmonary, hepatic, rheumatologic, autoimmune, or renal disease based on history, physical examination, and/or laboratory studies.
* Any other condition that, in the opinion of the investigator, would jeopardize the safety or rights of a subject participating in the trial, or would render the subject unable to comply with the protocol.
* History of a severe allergic reaction or anaphylaxis.
* Any known immunodeficiency syndrome.
* HIV infection, by screening and confirmatory assays (performed within 14 days of ZIKV challenge).
* Hepatitis C virus (HCV) infection, by screening and confirmatory assays.
* Hepatitis B virus (HBV) infection, by Hepatitis B surface antigen (HBsAg) screening.
* Current use of anticoagulant medications (this does not include anti-platelet medication such as aspirin or non-steroidal anti-inflammatory medications).
* Use of corticosteroids (excluding topical, inhaled, or nasal) or immunosuppressive drugs within 28 days prior to or following challenge. An immunosuppressive dose of corticosteroids is defined as ≥ 10 mg of a prednisone equivalent per day for ≥14 days.
* Receipt of a live vaccine within 28 days or an inactivated or subprotein vaccine within the 14 days prior to inoculation or anticipated receipt of any vaccine during the 28 days following inoculation with the exception of the inactivated influenza vaccine and COVID-19 vaccines either licensed or under EUA which can be given at any time, however all effort will be made to avoid giving influenza and COVID-19 vaccines within the above windows.
* Asplenia.
* Receipt of blood products within the past 6 months, including transfusions or immunoglobulin, or anticipated receipt of any blood products or immunoglobulin during the 28 days following challenge.
* Anticipated receipt of any other investigational agent in the 28 days before or after challenge.
* Definite plans to travel to a dengue-endemic area during the remainder of the study.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 26 (Estimated)
Dates: Start 2024-09-24 (Actual); Primary Completion 2025-09 (Estimated); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
Incidence, magnitude, and duration of infectious ZIKV-SJRP/2016-184 recovered from serum following administration of ZIKV-SJRP/2016-184 in subjects who received TV003 | Through 180 days post challenge
  Compared to historical controls
Incidence, magnitude, and duration of infectious ZIKV-SJRP/2016-184 recovered from serum following administration of ZIKV-SJRP/2016-184 in ZIKV-exposed subjects | Through 180 days post challenge
  Compared to historical controls
Proportion of subjects who received TV003 who develop clinical signs/symptoms of Zika infection | Through 180 days post challenge
  Compared to historical controls
Proportion of subjects who were previously infected with ZIKV who develop clinical signs/symptoms of Zika infection | Through 180 days post challenge
  Compared to historical controls
Frequency of immediate, systemic, and local adverse events (AEs) following vaccination with TV003 | Through 28 days post vaccination
Frequency of immediate, systemic, and local AEs following inoculation with ZIKV-SJRP/2016-184 | Through 28 days post challenge

SECONDARY OUTCOMES:
Incidence, magnitude, and duration of ZIKV viremia induced by administering 10^2 PFU of ZIKV-SJRP/2016-184 in subjects who received TV003 | Through 6 months post challenge
  Measured by quantitative polymerase chain reaction (PCR) induced, compared to historical controls.
Incidence, magnitude, and duration of ZIKV viremia induced by administering 10^2 PFU of ZIKV-SJRP/2016-184 in previously ZIKV-exposed subjects | Through 6 months post challenge
  Measured by quantitative PCR induced, compared to historical controls.
Number of TV003 vaccinees infected with DENV-1, DENV-2, DENV-3, and DENV-4 following administration of TV003 | Through 270 days post vaccination
  Infection is defined as recovery of vaccine virus from the blood or serum of a subject and/or by seropositivity to DENV measured by quantitative PCR
Peak neutralizing antibody titer (NT) to DENV-1, DENV-2, DENV-3, and DENV-4 | Through 90 days post vaccination
  Measured by the NT50 at 28, 56, and 90 days after TV003 vaccination.
Peak NT to ZIKV-SJRP/2016-184 | Through 90 days post challenge
  Measured by NT50 at 0, 28, 56, and 90 days post-administration of ZIKV-SJRP
Number of volunteers who become infected following primary ZIKV-SJRP administration | Through 16 days post challenge
Peak NT50 against ZIKV following TV003 vaccination correlates with protection against ZIKV infection | Through 90 days post challenge
Evaluate boost in neutralizing antibody titers to DENV-1, DENV-2, DENV-3, and DENV-4 post-ZIKV challenge in subjects who received TV003 | Through 90 days post challenge
  Peak NT50 achieved through 90 days post-ZIKV challenge in TV003 recipients. A boost in antibody titer is defined as a ≥ 4-fold rise through 90 days post challenge compared with the titer just prior to ZIKV challenge.
Evaluate boost in neutralizing antibody titers to ZIKV post challenge in subjects with previous ZIKV infection | Through 90 days post-ZIKV challenge of previous ZIKV recipients
  Peak NT50 achieved through 90 days post-ZIKV challenge. A boost in antibody titer is defined as a ≥ 4-fold rise in peak ZIKV neutralizing antibody titer through 90 days post challenge compared with the ZIKV neutralizing antibody titer in serum collected just prior to ZIKV challenge.
Quantity and duration of ZIKV in blood, cervico-vaginal secretions and semen | Through 6 months post challenge
  Measured by culture (infectious virus) and by reverse transcriptase - PCR in all participants receiving ZIKV-SJRP/2016-184

CONTACTS AND LOCATIONS:
Overall Officials: Anna Durbin, M.D., Principal Investigator — Johns Hopkins Bloomberg School of Public Health
Locations (2):
- United States (2):
  - Center for Immunization Research, Johns Hopkins School of Public Health, Baltimore, Maryland
  - Center for Immunization Research, Baltimore, Maryland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Pierce KK, Durbin AP, Walsh MR, Carmolli M, Sabundayo BP, Dickson DM, Diehl SA, Whitehead SS, Kirkpatrick BD. TV005 dengue vaccine protects against dengue serotypes 2 and 3 in two controlled human infection studies. J Clin Invest. 2024 Feb 1;134(3):e173328. doi: 10.1172/JCI173328. PMID 37971871
- [Background] Durbin AP, Kirkpatrick BD, Pierce KK, Schmidt AC, Whitehead SS. Development and clinical evaluation of multiple investigational monovalent DENV vaccines to identify components for inclusion in a live attenuated tetravalent DENV vaccine. Vaccine. 2011 Sep 23;29(42):7242-50. doi: 10.1016/j.vaccine.2011.07.023. Epub 2011 Jul 21. PMID 21781997
- [Background] Kallas EG, Cintra MAT, Moreira JA, Patino EG, Braga PE, Tenorio JCV, Infante V, Palacios R, de Lacerda MVG, Batista Pereira D, da Fonseca AJ, Gurgel RQ, Coelho IC, Fontes CJF, Marques ETA, Romero GAS, Teixeira MM, Siqueira AM, Barral AMP, Boaventura VS, Ramos F, Elias Junior E, Cassio de Moraes J, Covas DT, Kalil J, Precioso AR, Whitehead SS, Esteves-Jaramillo A, Shekar T, Lee JJ, Macey J, Kelner SG, Coller BG, Boulos FC, Nogueira ML. Live, Attenuated, Tetravalent Butantan-Dengue Vaccine in Children and Adults. N Engl J Med. 2024 Feb 1;390(5):397-408. doi: 10.1056/NEJMoa2301790. PMID 38294972